CLINICAL TRIAL: NCT03332641
Title: A 12-week, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Citron(Citrus Junos Siebold ex Tanaka) Peel Extract on Improvement of Blood Cholesterol
Brief Title: Effect of Intake of Citron(Citrus Junos Siebold ex Tanaka) Peel Extract on Blood Cholesterol.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Yongsoon Park, Professor, Hanyang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HYI-17-060-1
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citron peel Extract (Experimental): Citron peel extract for 12 weeks
  Interventions: Dietary Supplement: Citron peel extract
- Placebo (Placebo Comparator): Placebo for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Citron peel extract — Citron peel extract for 12 weeks
  Arms: Citron peel Extract
Dietary Supplement: Placebo — Placebo for 12 weeks
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of Citron(Citrus Junos Siebold ex Tanaka) Peel Extract on improvement of Blood Cholesterol.

DETAILED DESCRIPTION:
This study was a 12 weeks, randomized, double-blind, placebo-controlled human trial. Twenty subjects were randomly divided into Citron(Citrus Junos Siebold ex Tanaka) Peel Extract or a placebo group. Blood cholesterol profiles before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-75 years with Total cholesterol 200-239 mg/dL

Exclusion Criteria:

* Lipid lowering agent within past 6 months
* Severe cardiovascular disease(Mvodardial infarction, stroke, etc)
* Renal disease(Heredity hyperlipidemia, Acute/Chronic renal failure, Nephrotic syndrome, ect)
* Cancer, Respiratory organ disease(Asthma, Chronic obstructive pulmonary disease)
* Diabetes mellitus
* Allergic or hypersensitive to any of the ingredients in the test products
* History of disease that could interfere with the test products or impede their absorption
* Under antipsychotic drugs therapy within past 2 months
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test by show the following results
* Pregnancy or breast feeding
* Not Contraception(except: Surgery for female infertility)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Changes of Cholesterol | 12 weeks
  Changes of Cholesterol were assessed before and after the intervention

SECONDARY OUTCOMES:
Changes of Lipid profile | 12 weeks
  Changes of Lipid profile were assessed before and after the intervention
Changes of Oxidized LDL | 12 weeks
  Changes of Oxidized LDL were assessed before and after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University, Seoul, South Korea